CLINICAL TRIAL: NCT02019823
Title: SMS-text Adherence Support (StAR*) Study, a Randomized Three-arm Open Parallel Group Trial to Evaluate the Effects of a Structured Programme of Hypertension Treatment Adherence Support Delivered Remotely Through SMS-text Messages on Blood Pressure at 12 Months as Compared With Usual Care.
Brief Title: Effectiveness of SMS-text Message Support for Patients With Hypertension to Improve Blood Pressure
Acronym: *StAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); EPSRC (Unknown); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMSBP; NHREC# 2868 (Registry Identifier: South African National Clinical Trials Register); 418/2011 (Other: University of Cape Town Human Subjects Research Ethics Committee); 141/2011 (Other: Western Cape Province Department of Health Research Committee)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension; SMS-text; mHealth
Keywords: SMS-text; mobile health; mHealth; treatment; adherence
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enhanced usual care (Active Comparator): In addition to usual care participants will receive the pre-randomisation "Welcome to the *StAR Study" SMS-text, post-randomisation they will received a "Happy Birthday" SMS-text on their date of birth and up to six additional SMS-text messages containing study specific information and thanking the participant for taking part in the study. Participants in the Enhanced Usual Care group will receive no more than one study specific SMS-text every two months.
  Interventions: Behavioral: Enhanced usual care
- Informational SMS-text (Experimental): In addition to enhanced usual care, participants allocated to the informational SMS-text support group will receive a series of text-messages covering the following areas:
  I. Medication pick-up reminders send 48 hours before scheduled medication pick-up date a) Participants who fail to pick-up medication within 3 days of scheduled pick-up date will be sent one further reminder SMS-text
  II. III. Clinic appointment reminder 48 hours before scheduled follow-up appointment
  a) Participants who fail to attend clinic appointment will be sent an additional SMS-text checking they are alright and inviting them to rebook their appointment via the clinic IV. Messages which support medication adherence (focused on organisation, memory, and habit) or provide hypertension related health information
  Interventions: Behavioral: Informational SMS-text; Behavioral: Enhanced usual care
- Interactive SMS-text (Experimental): In addition to enhanced usual care and informational SMS-text messages, SMS-text messages sent to participants in the interactive SMS-text group will contain a "prompt to respond" which will guide participants to additional SMS-text based resources.
  Interventions: Behavioral: Informational SMS-text; Behavioral: Interactive SMS-text; Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Informational SMS-text
  Arms: Informational SMS-text; Interactive SMS-text
Behavioral: Interactive SMS-text
  Arms: Interactive SMS-text
Behavioral: Enhanced usual care

SUMMARY:
General synopsis for SMS-text Adherence Support (*StAR) Study and associated preparatory and pilot work

Background: High blood pressure is an important risk factor for heart disease, stroke and chronic kidney disease. Clear evidence exists that for individuals with high blood pressure (hypertension) lowering blood pressure really reduces this risk. One of the critical factors in the long term control of blood pressure is the regular use of effective antihypertensive medications. In South Africa, poor treatment adherence (attending clinic, re-filling prescriptions, and regularly taking hypertension tablets) is known to be an important and alterable risk factor for uncontrolled high blood pressure and its complications (heart disease, stroke and chronic kidney disease). SMS-text messages have been shown to improve clinic attendance and medication adherence for some diseases (like HIV and TB) in other low-resource settings. It is not clear whether SMS-text messages to support treatment adherence have an effect on long-term blood pressure control. The acceptability, sustainability and scalability such technology also remains to be determined.

Aim: To investigate if a system of SMS-text messages to support treatment adherence is more effective than usual care for controlling high blood-pressure.

Objectives: The main objective is to test whether advice and support given by SMS-text, either by providing information (informational) or by allowing a two-way communication (interactive) improves control of blood pressure at one year compared to usual care.

Additional objectives include assessing whether the interventions have an effect on,

* Clinic attendance
* Prescription refill adherence
* Self-reported medication adherence
* Hypertension related illness or death
* Patient empowerment

Study design: Single centre randomized three-arm parallel group trial As it is not clear how best to support treatment adherence for people with hypertension we need to compare the different ways this might be done. Eligible patients who provide written consent will be put into one of three groups and then compared. The groups are selected by a computer which has no information about the individual (i.e. by chance). Participants in each group will get different types of SMS-text messages and these are compared.

Study interventions:

* Enhanced usual care In addition to their usual clinical care participants will receive the pre-randomisation "Welcome to the *StAR Study" SMS-text, a "Happy Birthday" SMS-text on their date of birth and up to six additional SMS-text messages containing study specific information and thanking the participant for taking part in the study.
* Informational SMS-text messages In addition to enhanced usual care, participants allocated to the informational SMS-text support group will receive semi-tailored structured adherence-support (including clinic appointment and medication pick-up reminders, medication adherence support and hypertension-related education.)
* Interactive SMS-text messages In addition to enhanced usual care and informational SMS-text messages, SMS-text messages sent to participants in the interactive SMS-text group will contain a "prompt to respond" which will guide participants to additional SMS-text based resources.

Outcome measures: The main outcome measure is mean blood pressure measured at one year. Additional outcomes include the proportion of participants with "controlled blood pressure" as well as measures of clinic attendance, prescription refill adherence, self-reported medication adherence, hypertension related illness or death, and patient empowerment.

DETAILED DESCRIPTION:
General synopsis for SMS-text Adherence Support (*StAR) Study and associated preparatory and pilot work

Background: High blood pressure is an important risk factor for heart disease, stroke and chronic kidney disease. Clear evidence exists that for individuals with high blood pressure (hypertension) lowering blood pressure really reduces this risk. One of the critical factors in the long term control of blood pressure is the regular use of effective antihypertensive medications. In South Africa, poor treatment adherence (attending clinic, re-filling prescriptions, and regularly taking hypertension tablets) is known to be an important and alterable risk factor for uncontrolled high blood pressure and its complications (heart disease, stroke and chronic kidney disease). SMS-text messages have been shown to improve clinic attendance and medication adherence for some diseases (like HIV and TB) in other low-resource settings. It is not clear whether SMS-text messages to support treatment adherence have an effect on long-term blood pressure control. The acceptability, sustainability and scalability such technology also remains to be determined.

Aim: To investigate if a system of SMS-text messages to support treatment adherence is more effective than usual care for controlling high blood-pressure.

Objectives: The main objective is to test whether advice and support given by SMS-text, either by providing information (informational) or by allowing a two-way communication (interactive) improves control of blood pressure at one year compared to usual care.

Additional objectives include assessing whether the interventions have an effect on,

* Clinic attendance
* Prescription refill adherence
* Self-reported medication adherence
* Hypertension related illness or death
* Patient empowerment

Study design: Single centre randomized three-arm parallel group trial As it is not clear how best to support treatment adherence for people with hypertension we need to compare the different ways this might be done. Eligible patients who provide written consent will be put into one of three groups and then compared. The groups are selected by a computer which has no information about the individual (i.e. by chance). Participants in each group will get different types of SMS-text messages and these are compared.

Study interventions:

* Enhanced usual care In addition to their usual clinical care participants will receive the pre-randomisation "Welcome to the *StAR Study" SMS-text, a "Happy Birthday" SMS-text on their date of birth and up to six additional SMS-text messages containing study specific information and thanking the participant for taking part in the study.
* Informational SMS-text messages In addition to enhanced usual care, participants allocated to the informational SMS-text support group will receive semi-tailored structured adherence-support (including clinic appointment and medication pick-up reminders, medication adherence support and hypertension-related education.)
* Interactive SMS-text messages In addition to enhanced usual care and informational SMS-text messages, SMS-text messages sent to participants in the interactive SMS-text group will contain a "prompt to respond" which will guide participants to additional SMS-text based resources.

Outcome measures: The main outcome measure is mean blood pressure measured at one year. Additional outcomes include the proportion of participants with "controlled blood pressure" as well as measures of clinic attendance, prescription refill adherence, self-reported medication adherence, hypertension related illness or death, and patient empowerment.

Participant recruitment:

Posters advertising the study and leaflets containing study information will be available in the general waiting areas of the health centre. Adult patients attending the medical outpatients department or one of the chronic disease clubs will be approached and invited to consider taking part in the study. Interested individuals will have the opportunity to ask trained research staff questions about the study and their participation. Information about the study will be available in English, isi-Xhosa, and Afrikaans. Individuals interested in participating will be asked a series of screening questions to assess their eligibility for inclusion in the study and will have their blood pressure measured as per the study protocol. Eligible participants who decline to participate will be asked for permission to access their clinical record to extract basic details (age, gender, medication, recent blood pressure). Copies of Participant Information Leaflets and posters in English can be found in Appendix B. Translated copies are available upon request.

Informed consent procedures:

Eligible individuals who agree to participate will be asked to complete a consent form. A copy of the completed form will be given to participants as part of their trial information pack. Copies of consent to participate forms in English can be found in Appendix B. Translated copies are available upon request.

Study assessments:

* Baseline We will ask standard questions about health and medical history, and measure blood pressure, weight and height. Any necessary blood tests will be done as per clinic protocols. A trained research assistant will review participant's clinical records.
* 6 months Participant contact details (particularly participant's primary mobile-telephone number) will be checked and if necessary up-dated and blood pressure will be measured.
* 12 months A trained research assistant will administer a final set of questionnaires, measure participant's blood pressure according to the trial protocol, and repeat basic clinical measurements including anthropometry. Clinical records will be reviewed to capture intervening clinical events and changes in medical management. Participants who do not attend the 12 month follow-up clinic appointment will be followed up, and if cause for non-attendance is hospital admission or death, then hospital records or death certificate data will be obtained.

End of the study:

The end of study is the date of the final 12-month follow-up clinic visit of the last participant. After this time study participants will be asked if they would like to receive SMS-text messages as per the provincial department of health protocol if it exists.

Privacy and confidentiality:

Participant's contact details (cellular phone number, address, etc), these will only be available to name senior research staff involved in the study. Details will not be shared with the clinic staff or with any other service provider unless permission to do so is expressly given by the participant once the study has concluded. Data will be captured using a combination of electronic data capture and paper case-report forms (CRFs). CRFs will be entered onto the trial database on the day of collection. The trial database will include checks for logic and consistency to be resolved by the local investigators. Data will be stored on a computer with individually assigned passwords and individually assigned levels of access. The trial database will include a full audit trail of any changes made. Randomisation codes will be separately stored and accessible only by the trial statistician. No personal data will be included in the trial database and participants will be identifiable only by a unique study number. All essential documents will be retained in a trial master file. Trial documentation will be archived and stored for seven years.

Potential for harm:

The measurements we propose to take including blood pressure, height, weight, and waist circumference are very safe and are regularly used in routine clinical care. We will be taking participant's blood pressure a few more times than is usually done in the clinic which could cause some discomfort. The potential for harm to patients as a result of the trial intervention is judged as low. The University maintains Public Liability and Professional Liability insurance which will operate in this respect.

Potential benefits to individual participants:

All study participants will receive SMS-text messages which they may find beneficial. Participants will have their blood pressure accurately measured on at least three occasions.

Rewards:

This study is not providing any rewards or compensation to participants. Study participants are not provided cell-phones or network airtime credit, however receiving SMS-texts or phone calls or sending please call me messages to the study are free.

Study funding:

This study is funded as part of a programme grant from the Wellcome Trust and EPSRC (Grant Number DFR RDV0).

Pilot and preparatory work prior to the starting the StAR* study:

The protocol also includes brief summaries of preparatory and pilot work that will be carried out to optimise the trial design and procedures prior to beginning the StAR* study (these "StAR* study development phase projects" can be found in section 11 of the study protocol).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension and are either currently receiving or are about to start blood pressure lowering medication
* Mean blood pressure at enrolment is < 175/105
* Aged 21 years or older
* Must have access to a cell-phone (shared access is allowed if access is daily and the phone owner agrees to participate)
* Must be able to use SMS-text (help by a partner is allowed for illiterate subjects, subjects with poor vision, or subjects who are learning disabled)
* Must be resident in the study area and must be expected to be resident for the duration of the study

Exclusion Criteria:

* Another member of the household has already been recruited into the trial
* If female, they are not pregnant or within three months post-partum by self-report
* They are not willing to give informed consent and take part in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1372 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 12-months from baseline
  The primary outcome is change in systolic blood pressure which we will analyse using a mixed-effects model on data collected at 6 and 12-months.

SECONDARY OUTCOMES:
Measured treatment adherence | 3-monthly intervals over 12-months of follow-up
  Treatment adherence is assessed by calculating the proportion of days covered from routinely collected prescribing and dispensing data obtained during the 12-month follow-up period.

OTHER OUTCOMES:
Proportion of participants with a systolic blood pressure < 140 mmHg and a diastolic blood pressure <90 mmHg | At 12-months
Hospital admissions for hypertension related illnesses | At 12-months
Self-reported health status | At 12-months
  EuroQol 5-Dimension and Visual Analogue Scale
Proportion of scheduled clinic appointments attended | At 12-months
Satisfaction with clinic services and care | At 12-months
  Assessed using 12 5-point Likert-scale items adapted from locally appropriate questionnaires developed to capture patient satisfaction with services.
Self-reported adherence to antihypertensive treatment | At 12-months
Basic knowledge about hypertension | At 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Tarassenko, MA, DPhil, FREng, FIET, Study Chair — University of Oxford; Andrew Farmer, DM FRCGP, Principal Investigator — University of Oxford; Naomi Levitt, MBChB, MD and FCP(SA)), Principal Investigator — University of Cape Town

REFERENCES:
- [Background] Bobrow K, Brennan T, Springer D, Levitt NS, Rayner B, Namane M, Yu LM, Tarassenko L, Farmer A. Efficacy of a text messaging (SMS) based intervention for adults with hypertension: protocol for the StAR (SMS Text-message Adherence suppoRt trial) randomised controlled trial. BMC Public Health. 2014 Jan 11;14:28. doi: 10.1186/1471-2458-14-28. PMID 24410738
- [Derived] Bobrow K, Farmer A, Cishe N, Nwagi N, Namane M, Brennan TP, Springer D, Tarassenko L, Levitt N. Using the Medical Research Council framework for development and evaluation of complex interventions in a low resource setting to develop a theory-based treatment support intervention delivered via SMS text message to improve blood pressure control. BMC Health Serv Res. 2018 Jan 23;18(1):33. doi: 10.1186/s12913-017-2808-9. PMID 29361934
- [Derived] Bobrow K, Farmer AJ, Springer D, Shanyinde M, Yu LM, Brennan T, Rayner B, Namane M, Steyn K, Tarassenko L, Levitt N. Mobile Phone Text Messages to Support Treatment Adherence in Adults With High Blood Pressure (SMS-Text Adherence Support [StAR]): A Single-Blind, Randomized Trial. Circulation. 2016 Feb 9;133(6):592-600. doi: 10.1161/CIRCULATIONAHA.115.017530. Epub 2016 Jan 14. PMID 26769742
- [Derived] Leon N, Surender R, Bobrow K, Muller J, Farmer A. Improving treatment adherence for blood pressure lowering via mobile phone SMS-messages in South Africa: a qualitative evaluation of the SMS-text Adherence SuppoRt (StAR) trial. BMC Fam Pract. 2015 Jul 3;16:80. doi: 10.1186/s12875-015-0289-7. PMID 26137844